CLINICAL TRIAL: NCT03388892
Title: A Randomized Controlled Trial of Drug-Eluting Balloon Angioplasty in Venous Anastomotic Stenosis of Dialysis Arteriovenous Graft
Brief Title: Drug-Eluting Balloon in Arteriovenous Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-065-F
Record Dates: First submitted 2015-12-02; First posted 2018-01-03 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Kidney Failure, Chronic; Angioplasty; Dialysis
Keywords: Angioplasty; Drug Eluting Balloon; Arteriovenous Graft
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-Eluting Balloon (Experimental): PTA with DEB at venous anastomotic stenosis of AVG
  Interventions: Device: paclitaxel-coated balloon, IN. PACT(Invatec-Medtronic, Brescia, Italy)
- Plain Balloon (Active Comparator): PTA with PCB at venous anastomotic stenosis of AVG
  Interventions: Device: Plain Balloon

INTERVENTIONS:
Device: paclitaxel-coated balloon, IN. PACT(Invatec-Medtronic, Brescia, Italy) — Arteriovenous graft (AVG) dysfunction or acute thrombosis is mainly caused by neointimal hyperplasia. Although endovascular intervention, such as percutaneous transluminal angioplasty (PTA), catheter-based directed thrombolysis with urokinase, mechanical thrombectomy with percutaneous thrombolytic device or even if graft stenting, can salvage the hemodialysis access, the long-term primary and secondary patent rate don't improve due to repeated restenosis from neointimal hyperplasia. Drug eluting balloon is used in reducing neointimal hypoplasia in patients with coronary in-stent restenosis and it's also effective in restenosis of peripheral arterial diseases. It's reasonable to hypothesize that PTA with PCB at venous anastomotic stenosis of AVG could prolong the patency and reduce the acute thrombosis rate.
  Arms: Drug-Eluting Balloon
Device: Plain Balloon — Traditional Plain Balloon was used to dilate the venous anastomotic stenosis of arteriovenous graft (AVG) as the usual intervention
  Arms: Plain Balloon

SUMMARY:
The investigators' study aims is to evaluate the safety and efficacy of percutaneous transluminal angioplasty (PTA) with paclitaxel-coated balloon (PCB) at venous anastomotic stenosis of arteriovenous graft (AVG) in patients with hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 90 years
2. Patients under hemodialysis via prosthetic arteriovenous graft in the arm
3. Vascular access was created for more than 30 days and used at least one successful session
4. Clinical failure for hemodialysis due to higher venous pressure or lower arterial flow
5. Angiography proved venous anastomotic stenosis ≥50% (the entire lesion of venous anastomotic stenosis will be extended into AVG no more than 2cm and naive vein no more than 7 cm). There was no other obvious stenosis.
6. Reference diameter of venous anastomosis within 7 mm

Exclusion Criteria:

1. Patient could not write informed consent
2. Being unwilling or unable to return for follow-up visits or reason to believe that adherence to follow-up visits would be irregular
3. Current or scheduled enrollment in other, conflicting studies.
4. Acute thrombosis in the past 3 months
5. Central venous stenosis
6. Concomitant disease (e.g., terminal cancer) or other medical condition likely to result in death within 6 months
7. A blood coagulation disorder
8. Sepsis or infected arteriovenous access graft
9. A contraindication to the use of contrast medium
10. Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
patent rate in percentage after PTA | 1 year
  Late luminal loss in patients was evaluated by quantitative angiography after PTA and intravascular ultrasound (IVUS) up to 12 months after PTA. Late luminal loss is defined as the difference between the minimal lumen diameter in percentage and the late luminal loss less than 50% was defined as patency.

SECONDARY OUTCOMES:
The incidence of angiography-guided binary restenosis rate (≥50% of the diameter of the reference-vessel) | 1 year
  Measure the stenotic percentage every 2 months up to 1 year for angiography
The incidence of IVUS-guided binary restenosis rate (≥50% of the diameter of the reference-vessel) | 1 year
  Measure the stenotic percentage 1, 6, 12 months for IVUS
Change of AVG flow in liter per minute | 1 year
  measure the AVG flow and pressure before PTA, 1 week and every 2 months up to 1 year after PTA
Change of AVG pressure in mmHg | 1 year
  measure the AVG flow and pressure before PTA, 1 week and every 2 months up to 1 year after PTA
Time interval of patent AVG after PTA | 1 year
  Patent AVG was defined as luminal loss less than 50%
The rate of AVG failure at 6 months and 12 months | 1 year
  AVG failure was defined as AVG thrombosis, AVG re-intervention

OTHER OUTCOMES:
Paclitaxel-coated balloon safety | 1 year
  Record complications of paclitaxel-coated balloon such as graft failure and vessel dissection or rupture.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

REFERENCES:
- [Derived] Liao MT, Lee CP, Lin TT, Jong CB, Chen TY, Lin L, Hsieh MY, Lin MS, Chie WC, Wu CC. A randomized controlled trial of drug-coated balloon angioplasty in venous anastomotic stenosis of dialysis arteriovenous grafts. J Vasc Surg. 2020 Jun;71(6):1994-2003. doi: 10.1016/j.jvs.2019.07.090. Epub 2019 Oct 11. PMID 31611105